CLINICAL TRIAL: NCT01111578
Title: Evaluation of a New Enteral Feeding Tube for the Measurement of Esophageal and Gastric Pressure
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, MD, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico
Other Study IDs: 17610
Record Dates: First submitted 2010-04-12; First posted 2010-04-27 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-04

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New enteral feeding tube
  Interventions: Device: Enteral feeding tube

INTERVENTIONS:
Device: Enteral feeding tube — The esophageal and gastric pressure, measured with this new device, will be recorded and compared with those ones measured with a standard esophageal catheter

SUMMARY:
Investigators aim to evaluate the accuracy in the measurement of the esophageal and gastric pressure of a new enteral feeding tube

ELIGIBILITY:
Inclusion Criteria:

* Requiring the placement of an enteral feeding tube

Exclusion Criteria:

* esophageal ulcers
* severe coagulophaty
* thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to a general and post-operative intensive care unit and who, for clinical reasons, need the placement of an enteral feeding tube
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of the measurement of the esophageal and gastric pressure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Fondazione IRRCS Ca' Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI, Italy